CLINICAL TRIAL: NCT06962709
Title: Comparing the Anesthetic Effect of Warmed Lidocaine to Room Temperature Lidocaine When Applied Topically for Intravitreal Injections
Brief Title: Studying Warmed Lidocaine for Increased Analgesic Effect During Intravitreal Injections
Acronym: WarmLido
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Balaji (Other)
Responsible Party: Sponsor-Investigator, Balaji, Investigator, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2090898
Record Dates: First submitted 2025-02-24; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Pain Intensity Assessment; Pain Management
Keywords: warmed lidocaine; intravitreal injections
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients receiving warmed lidocaine (Experimental): Patients receive lidocaine jelly that has been warmed before they receive an intravitreal injection.
  Interventions: Other: Warmed lidocaine
- Patients receiving room temperature lidocaine (No Intervention): Patients receive room temperature lidocaine before intravitreal injection

INTERVENTIONS:
Other: Warmed lidocaine — Lidocaine warmed to 98 F
  Arms: Patients receiving warmed lidocaine

SUMMARY:
Investigating whether warmed lidocaine increases analgesic effect for intravitreal injections

ELIGIBILITY:
Inclusion Criteria:

* Receiving intravitreal injection for any indication

Exclusion Criteria:

* Previous participant in study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain Rating | immediately after the intervention
  The level of pain associated with intravitreal injection as marked by patient on 10cm line.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital - Mason Eye Clinic, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No